CLINICAL TRIAL: NCT04148365
Title: Medication Compliance in the Paediatric Uveitis Population Reported by the Patients and Parents
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 257448; B00751 (Other: Manchester University NHS Foundation Trust)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Uveitis
Keywords: Paediatrics
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric Uveitis: Patients with Uveitis below the age of 18 years.

SUMMARY:
Little is known about eye drop regime adherence in the paediatric population. In particular, no previous research has investigated this in the paediatric uveitis population, a group who can require doses up to six times daily, and at frequencies that change month to month. The aim of the study is to quantify the range of adherence to eye drop medication, and to investigate some of the reasons for non-compliance in a child specific study. By learning more about compliance, this will help create treatments that are better suited to children.

The study will recruit 50 children receiving eye drop treatment. After an interval of 1 week or more the children and their parents will be asked to complete a questionnaire about the frequency of the drops prescribed, and the frequency that they have used over the last interval. It will also ask questions about difficulties encountered administering the drops.

Changes in eye drop bottle weight will be measured during the interval and the result compared.

The information gathered from the questionnaires will be used to compare reports of adherence between the parent and child, the child's age and the bottle weight. The reasons reported for difficulties with adherence will also be reported. This is a preliminary investigatory study to identify whether an issue with medication non-adherence exists. The findings will be used to tailor further research into this area.

DETAILED DESCRIPTION:
Purpose This study aims to provide new information about compliance with medications amongst children and adolescents in an outpatient Ophthalmic setting.

Previous studies have demonstrated in other conditions that adherence to eye drop regimes is extremely varied (50% to 90% of prescribed drops (Tan 2005)) in a range of paediatric conditions including myopia, amblyopia, herpes simplex keratitis, allergic conjunctivitis. There has not been any research into eye drop adherence in the paediatric uveitis population. Previous enquiries into quality of life in JIA have not included questions about drop adherence, frequency of flare ups or drop side effects (van Dijkhuizen 2018). Although this condition is not common, the prevalence of paediatric uveitis is 27.9 per 100,000 (Päivönsalo-Hietanen 2000), it has severe sight threatening complications despite modern treatment. The burden of disease can be substantial due to eye drops up to six times daily and weekly appointments during active episodes, as well as surveillance every 3-4 months in between flares.

There are certain issues that are specific to uveitis which require investigation. These include the high frequency of steroid drops, changes in frequency on a week by week basis, and the fact that it is an asymptomatic condition in the early stages. Other studies reporting drop adherence in the paediatric population are limited because definitions of adherence and its measurement is inconsistent, and often not the primary outcome of a study. Parents and clinicians have expressed concerns about how achievable very frequent dosing is. If a threshold above which eye drop adherence becomes very unreliable exists, for instance more than four times each day, then clinicans could adjust treatment regimes to reflect this. This may encourage clinicans to be able to confidently advocate moving on to alternative therapies, such as biological treatment rather than increasing drop frequency.

By measuring and understanding medication adherence in the paediatric and adolescent population helps design interventions to improve compliance and assess their success. Evidence of paediatric specific issues may also lead to the development of age adapted formulations or trial of existing products in novel ways, for instance slow release steroid inserts following paediatric cataract surgery (SY Lee 2002).

Design Treatment will not be impacted by the study. There is no randomisation. Compliance may be impacted by awareness of being involved in a study. This is a major limitation of the study.

However previous studies have been conducted investigating compliance and their finding have been held to be valid.

A effort has been made in the design of PIS to provide patients with information about the study while limiting the impression that their medication compliance is under scrutiny. Additional vague questions have been added to the questionnaire to obscure the focus of the questions.

ELIGIBILITY:
Inclusion Criteria:

* Any child attending the Paediatric Ophthalmology Department Uveitis Clinic who is receiving eye drop treatment.
* Children with a diagnosis of uveitis receiving eye drop treatment between 0-18 years of age at the time of recruitment.

Exclusion Criteria:

* Children with follow up more than 3 months after the first meeting and consent will subsequently be excluded.
* At present the study does not have sufficient funding for translators. Potential participants that do not speak sufficient English to understand and respond to the questionnaire will be excluded. We hope to obtain additional funding following this preliminary research. A priority of any further work will be to provide translators and achieve a more inclusive approach.
* Children not accompanied by a person with parental responsibility will be excluded if they cannot provide their own consent.

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric uveitis population who attend Paediatric Ophthalmology Department Uveitis Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Frequency of reported medication errors (missed doses) among paediatric uveitis population. | 01/07/2020
  to determine what level of compliance with eye drop regimes currently exists in the paediatric uveitis population.

SECONDARY OUTCOMES:
What factors effect adherence to eye drop regimes? Including the frequency of eye drops and who administers the eye drops. | 01/07/2020
  Idenifying factors affecting adherence to taking eye drops
Does the age of the child influence compliance? | 01/07/2020
  What age is best compliant with eye drops
In children that are old enough to report drop use, is reported compliance comparable between child and parent? | 01/07/2020
  Parent and child compliancy

CONTACTS AND LOCATIONS:
Overall Officials: Jane Ashworth, Principal Investigator — Consultant Peadiatric Ophthalmologist
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No